CLINICAL TRIAL: NCT06366646
Title: Impact of Competency-Based Intervention on Leadership Effectiveness of Head Nurses in Teaching Hospitals
Brief Title: Competency-based Intervention for Head Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Nagah Abd El-Fattah Mohamed Aly, Assistant professor of Nursing administration, Matrouh University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 035901
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Intervention; Knowledge, Attitudes, Practice
Keywords: leadership; Competency; Effectiveness; Intervention; Program; Head nurses
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design
Who Masked: Participant
Masking Description: A quasi-experimental design utilized one group for pre-, post, and follow-up intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group of head nurses (Other): Head nurses received competency-based intervention
  Interventions: Other: Competency-based intervention
- group of assistant head nurses (Other): assistant head nurses received competency-based intervention
  Interventions: Other: Competency-based intervention

INTERVENTIONS:
Other: Competency-based intervention — 90 head nurses and their assistants received the competency-based intervention program

SUMMARY:
Head nurses have a crucial leadership role in managing their units and providing high-quality and safe nursing care. Head nurse leadership competency and effectiveness are very essential to manage nursing care practices and management activities in their hospitals. Development leadership competency intervention programs would improve the head nurse's competency and effectiveness.

DETAILED DESCRIPTION:
Head nurses have a crucial leadership role in managing their units and providing high-quality and safe nursing care. Head nurse leadership competency and effectiveness are very essential to manage nursing care practices and management activities in their hospitals. Development leadership competency intervention programs would improve the head nurse's competency and effectiveness. This study aimed to evaluate the impact of the leadership competency intervention program on the leadership effectiveness of head nurses

ELIGIBILITY:
Inclusion Criteria:

* Head nurses

  * willing to participate in the study
  * work in general wards and toxicology, intensive and critical care units
  * Sign a consent

Exclusion Criteria:

* Head nurses

  * work in outpatient units
  * Did not sign a consent
  * Absent from training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure head nurses' knowledge of leadership competency | one month
  Head nurses' Knowledge of competency as assessed using five Likert scales (ranging from (1) not essential to (5) extremely essential with each statement).
Questionnaire to measure head nurses' ability to use leadership competency | one month
  Head nurses perceived their ability to use leadership competency as assessed using five Likert scales (from 1 = never / no to 5 = always / yes).
Questionnaire to measure leadership effectiveness | one month
  Leadership effectiveness as assessed using a five Likert scale (1= strongly disagree and 5= strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Nagah Abd El-Fattah Mohamed Aly, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University, Egypt; Wael M. Lotfy, Ph.D, Study Director — Faculty of Nursing, Matrouh University, Egypt; Safaa M. El-Shanawany, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Maha Ghanem, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Elham Abd El KaderFayad, Ph.D, Study Chair — Psychatric Nursing and Mental health , Faculty of Nursing, Alexandria University, Egypt
Locations (1):
- Faculty of Nursing, Matrouh University, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No